CLINICAL TRIAL: NCT02144688
Title: CTNPT 015 - Pilot Project to Implement a Step-wise Investigation That Includes Cerebrospinal (CSF) Analysis as a Standard of Care for HIV+ Individuals With Cognitive Symptoms
Brief Title: COMO: Cognition Study With HIV+ Patients (CTNPT 015)
Acronym: COMO
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: In 14 participants who had LP, very low level viremia was found in only 1
Sponsor: Marie-Josée Brouillette (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government); CIHR Canadian HIV Trials Network (Network)
Responsible Party: Sponsor-Investigator, Marie-Josée Brouillette, Associate Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTNPT 015; NCT01848678 (obsolete NCT alias)
Record Dates: First submitted 2014-03-29; First posted 2014-05-22 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: HIV - Human Immunodeficiency Virus; Cognitive Symptoms
Keywords: Human Immunodeficiency Virus; HIV; Cognitive symptoms; Cognitive evaluation; Neuropsychological testing; Quality of life; Anxiety; Viral load; Antiretroviral; Cerebrospinal fluid; Lumbar puncture; Magnetic resonance imaging; MRI
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Neurobehavioral Manifestations; Anxiety Disorders | interventions — Anti-Retroviral Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Change in ARVs to improve cognition (Experimental): Change in ARVs to improve cognition: Personalized change in antiretrovirals will be based on CSF analysis
  Interventions: Drug: Change in antiretrovirals

INTERVENTIONS:
Drug: Change in antiretrovirals — Change in ARVs to improve cognition: Personalized change in antiretrovirals will be based on CSF analysis

SUMMARY:
The purpose of this study is to contribute evidence towards the potential to improve cognition in HIV+ individuals experiencing cognitive decline through personalized change in antiretroviral (ARV) medication. To that end, following a comprehensive evaluation to identify confounding clinical conditions, study participants will undergo a lumbar puncture to: (i) measure viral load (at 2 copies/ml); (ii) identify Cerebrospinal Fluid (CSF) genotype and tropism; and (iii) measure concentration of antiretroviral agents. When indicated from the CSF analysis, a personalized change in ARV will be implemented. Cognition will be measured in all at study entry and 6 months later.

ELIGIBILITY:
Inclusion Criteria:

* are 18 years and older
* have the capacity to give informed consent as determined by the research nurse
* have unexplained cognitive decline (reported either by the patient or an outside informant)
* have been on a stable ART regimen for > 6 months
* have an undetectable viral load in plasma for at least 6 months (a single blip of ≤ 150 copies/mL will be accepted)
* have not had a change in medications that could potentially interfere with cognition in the past 4 months

Exclusion Criteria:

* detectable VL in the plasma
* past history of dementia
* past history of Central Nervous System opportunistic infection or stroke
* current substance abuse ( as per DSM-IV criteria) other than cigarettes
* coagulopathy
* thrombocytopenia
* use of Coumadin
* intra-cranial hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Changes in neurocognitive functioning over 6 months | 6 months
  Cognition will be assessed at study entry and 6 months with the following tests: Letter Fluency, Category Fluency, Letter-Number Sequencing, Digit-Symbol, Symbol Search, Grooved Pegboard, Hopkins Verbal Learning Test-Revised, Stroop, Brief Visuospatial Memory Test-Revised, Tower of London, Trail Making Test A and B, Spatial Span, Montreal Cognitive Assessment (MoCA), and a brief computerized battery of tests (B-CAM).

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Josée Brouillette, MD, FRCPC, Principal Investigator — Montreal Chest Institute - Chronic Viral Illness Service - McGill University Health Centre (MUHC)
Locations (1):
- Montreal Chest Institute - Chronic Viral Illness Service - McGill University Health Centre (MUHC), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Antinori A, Arendt G, Becker JT, Brew BJ, Byrd DA, Cherner M, Clifford DB, Cinque P, Epstein LG, Goodkin K, Gisslen M, Grant I, Heaton RK, Joseph J, Marder K, Marra CM, McArthur JC, Nunn M, Price RW, Pulliam L, Robertson KR, Sacktor N, Valcour V, Wojna VE. Updated research nosology for HIV-associated neurocognitive disorders. Neurology. 2007 Oct 30;69(18):1789-99. doi: 10.1212/01.WNL.0000287431.88658.8b. Epub 2007 Oct 3. PMID 17914061
- [Background] Morrison NE, Collins FM. Immunogenicity of an aerogenic BCG vaccine in T-cell-depleted and normal mice. Infect Immun. 1975 May;11(5):1110-21. doi: 10.1128/iai.11.5.1110-1121.1975. PMID 123519
- [Background] Becker JT, Lopez OL, Dew MA, Aizenstein HJ. Prevalence of cognitive disorders differs as a function of age in HIV virus infection. AIDS. 2004 Jan 1;18 Suppl 1:S11-8. PMID 15075493
- [Background] Canestri A, Lescure FX, Jaureguiberry S, Moulignier A, Amiel C, Marcelin AG, Peytavin G, Tubiana R, Pialoux G, Katlama C. Discordance between cerebral spinal fluid and plasma HIV replication in patients with neurological symptoms who are receiving suppressive antiretroviral therapy. Clin Infect Dis. 2010 Mar 1;50(5):773-8. doi: 10.1086/650538. PMID 20100092
- [Background] Carey CL, Woods SP, Gonzalez R, Conover E, Marcotte TD, Grant I, Heaton RK; HNRC Group. Predictive validity of global deficit scores in detecting neuropsychological impairment in HIV infection. J Clin Exp Neuropsychol. 2004 May;26(3):307-19. doi: 10.1080/13803390490510031. PMID 15512922
- [Background] Cherner M, Ellis RJ, Lazzaretto D, Young C, Mindt MR, Atkinson JH, Grant I, Heaton RK; HIV Neurobehavioral Research Center Group. Effects of HIV-1 infection and aging on neurobehavioral functioning: preliminary findings. AIDS. 2004 Jan 1;18 Suppl 1:S27-34. PMID 15075495
- [Background] Cysique LA, Vaida F, Letendre S, Gibson S, Cherner M, Woods SP, McCutchan JA, Heaton RK, Ellis RJ. Dynamics of cognitive change in impaired HIV-positive patients initiating antiretroviral therapy. Neurology. 2009 Aug 4;73(5):342-8. doi: 10.1212/WNL.0b013e3181ab2b3b. Epub 2009 May 27. PMID 19474412
- [Background] Cysique LA, Brew BJ. Neuropsychological functioning and antiretroviral treatment in HIV/AIDS: a review. Neuropsychol Rev. 2009 Jun;19(2):169-85. doi: 10.1007/s11065-009-9092-3. Epub 2009 May 9. PMID 19424802
- [Background] Cysique LA, Maruff P, Brew BJ. Variable benefit in neuropsychological function in HIV-infected HAART-treated patients. Neurology. 2006 May 9;66(9):1447-50. doi: 10.1212/01.wnl.0000210477.63851.d3. PMID 16682686
- [Background] De Luca A, Ciancio BC, Larussa D, Murri R, Cingolani A, Rizzo MG, Giancola ML, Ammassari A, Ortona L. Correlates of independent HIV-1 replication in the CNS and of its control by antiretrovirals. Neurology. 2002 Aug 13;59(3):342-7. doi: 10.1212/wnl.59.3.342. PMID 12177366
- [Background] Ellis RJ, Moore DJ, Childers ME, Letendre S, McCutchan JA, Wolfson T, Spector SA, Hsia K, Heaton RK, Grant I. Progression to neuropsychological impairment in human immunodeficiency virus infection predicted by elevated cerebrospinal fluid levels of human immunodeficiency virus RNA. Arch Neurol. 2002 Jun;59(6):923-8. doi: 10.1001/archneur.59.6.923. PMID 12056927
- [Background] Florkowski CM. Sensitivity, specificity, receiver-operating characteristic (ROC) curves and likelihood ratios: communicating the performance of diagnostic tests. Clin Biochem Rev. 2008 Aug;29 Suppl 1(Suppl 1):S83-7. PMID 18852864
- [Background] Hardy DJ, Vance DE. The neuropsychology of HIV/AIDS in older adults. Neuropsychol Rev. 2009 Jun;19(2):263-72. doi: 10.1007/s11065-009-9087-0. Epub 2009 Feb 27. PMID 19247836
- [Background] McCutchan JA, Wu JW, Robertson K, Koletar SL, Ellis RJ, Cohn S, Taylor M, Woods S, Heaton R, Currier J, Williams PL. HIV suppression by HAART preserves cognitive function in advanced, immune-reconstituted AIDS patients. AIDS. 2007 May 31;21(9):1109-17. doi: 10.1097/QAD.0b013e3280ef6acd. PMID 17502721
- [Background] Jones RN, Gallo JJ. Dimensions of the Mini-Mental State Examination among community dwelling older adults. Psychol Med. 2000 May;30(3):605-18. doi: 10.1017/s0033291799001853. PMID 10883716
- [Background] Koski L, Xie H, Finch L. Measuring cognition in a geriatric outpatient clinic: Rasch analysis of the Montreal Cognitive Assessment. J Geriatr Psychiatry Neurol. 2009 Sep;22(3):151-60. doi: 10.1177/0891988709332944. Epub 2009 Mar 23. PMID 19307324
- [Background] Letendre S, Marquie-Beck J, Capparelli E, Best B, Clifford D, Collier AC, Gelman BB, McArthur JC, McCutchan JA, Morgello S, Simpson D, Grant I, Ellis RJ; CHARTER Group. Validation of the CNS Penetration-Effectiveness rank for quantifying antiretroviral penetration into the central nervous system. Arch Neurol. 2008 Jan;65(1):65-70. doi: 10.1001/archneurol.2007.31. PMID 18195140
- [Background] Letendre SL, McCutchan JA, Childers ME, Woods SP, Lazzaretto D, Heaton RK, Grant I, Ellis RJ; HNRC Group. Enhancing antiretroviral therapy for human immunodeficiency virus cognitive disorders. Ann Neurol. 2004 Sep;56(3):416-23. doi: 10.1002/ana.20198. PMID 15349869
- [Background] Marra CM, Lockhart D, Zunt JR, Perrin M, Coombs RW, Collier AC. Changes in CSF and plasma HIV-1 RNA and cognition after starting potent antiretroviral therapy. Neurology. 2003 Apr 22;60(8):1388-90. doi: 10.1212/01.wnl.0000058768.73358.1a. PMID 12707454
- [Background] Marra CM, Zhao Y, Clifford DB, Letendre S, Evans S, Henry K, Ellis RJ, Rodriguez B, Coombs RW, Schifitto G, McArthur JC, Robertson K; AIDS Clinical Trials Group 736 Study Team. Impact of combination antiretroviral therapy on cerebrospinal fluid HIV RNA and neurocognitive performance. AIDS. 2009 Jul 17;23(11):1359-66. doi: 10.1097/QAD.0b013e32832c4152. PMID 19424052
- [Background] Nath A, Sacktor N. Influence of highly active antiretroviral therapy on persistence of HIV in the central nervous system. Curr Opin Neurol. 2006 Aug;19(4):358-61. doi: 10.1097/01.wco.0000236614.51592.ca. PMID 16914973
- [Background] Nilsson C, Stahlberg F, Thomsen C, Henriksen O, Herning M, Owman C. Circadian variation in human cerebrospinal fluid production measured by magnetic resonance imaging. Am J Physiol. 1992 Jan;262(1 Pt 2):R20-4. doi: 10.1152/ajpregu.1992.262.1.R20. PMID 1733335
- [Background] Pilcher CD, Shugars DC, Fiscus SA, Miller WC, Menezes P, Giner J, Dean B, Robertson K, Hart CE, Lennox JL, Eron JJ Jr, Hicks CB. HIV in body fluids during primary HIV infection: implications for pathogenesis, treatment and public health. AIDS. 2001 May 4;15(7):837-45. doi: 10.1097/00002030-200105040-00004. PMID 11399956
- [Background] Price RW, Yiannoutsos CT, Clifford DB, Zaborski L, Tselis A, Sidtis JJ, Cohen B, Hall CD, Erice A, Henry K. Neurological outcomes in late HIV infection: adverse impact of neurological impairment on survival and protective effect of antiviral therapy. AIDS Clinical Trial Group and Neurological AIDS Research Consortium study team. AIDS. 1999 Sep 10;13(13):1677-85. doi: 10.1097/00002030-199909100-00011. PMID 10509569
- [Background] Robertson KR, Smurzynski M, Parsons TD, Wu K, Bosch RJ, Wu J, McArthur JC, Collier AC, Evans SR, Ellis RJ. The prevalence and incidence of neurocognitive impairment in the HAART era. AIDS. 2007 Sep 12;21(14):1915-21. doi: 10.1097/QAD.0b013e32828e4e27. PMID 17721099
- [Background] Robertson KR, Robertson WT, Ford S, Watson D, Fiscus S, Harp AG, Hall CD. Highly active antiretroviral therapy improves neurocognitive functioning. J Acquir Immune Defic Syndr. 2004 May 1;36(1):562-6. doi: 10.1097/00126334-200405010-00003. PMID 15097298
- [Background] Schultz-Larsen K, Kreiner S, Lomholt RK. Mini-Mental Status Examination: mixed Rasch model item analysis derived two different cognitive dimensions of the MMSE. J Clin Epidemiol. 2007 Mar;60(3):268-79. doi: 10.1016/j.jclinepi.2006.06.007. Epub 2006 Aug 10. PMID 17292021
- [Background] Valcour V, Shikuma C, Shiramizu B, Watters M, Poff P, Selnes O, Holck P, Grove J, Sacktor N. Higher frequency of dementia in older HIV-1 individuals: the Hawaii Aging with HIV-1 Cohort. Neurology. 2004 Sep 14;63(5):822-7. doi: 10.1212/01.wnl.0000134665.58343.8d. PMID 15365130
- [Background] Valcour V, Paul R. HIV infection and dementia in older adults. Clin Infect Dis. 2006 May 15;42(10):1449-54. doi: 10.1086/503565. Epub 2006 Apr 13. PMID 16619159
- [Background] Wouters H, van Gool WA, Schmand B, Lindeboom R. Revising the ADAS-cog for a more accurate assessment of cognitive impairment. Alzheimer Dis Assoc Disord. 2008 Jul-Sep;22(3):236-44. doi: 10.1097/WAD.0b013e318174f8b9. PMID 18580585